CLINICAL TRIAL: NCT07298811
Title: Preliminary Clinical Study of the Effectiveness and Safety of Ocular Surface Microbiota Transplantation in the Treatment of Dry Eye Disease: a Randomized, Single-blind,-Controlled Trial.
Brief Title: Preliminary Clinical Study of the Effectiveness and Safety of Ocular Surface Microbiota Transplantation in the Treatment of Dry Eye Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifeng Yu, Associate Chief Physician, Ph.D., Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT-I-2025-081
Record Dates: First submitted 2025-11-23; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye
Keywords: dry eye; ocular surface diseases; Microbiota transplantation
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplant group (Active Comparator): Transplant operation to dry eye patients
  Interventions: Biological: Ocular surface microbiota transplantation
- Placebo group (Placebo Comparator): Fake transplantation to dry eye patients
  Interventions: Biological: Placebo Group

INTERVENTIONS:
Biological: Ocular surface microbiota transplantation — Ocular surface microbiota transplantation
  Arms: Transplant group
Biological: Placebo Group — Fake transplant operation
  Arms: Placebo group

SUMMARY:
Evaluate the efficacy and safety of ocular surface microbiota transplantation as an adjunctive therapy for dry eye, and explore its impact on the structure of the ocular surface microbiota.

DETAILED DESCRIPTION:
Evaluate the efficacy and safety of ocular surface microbiota transplantation as an adjunctive therapy for dry eye, and explore its impact on the structure of the ocular surface microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Dry Eye Patient Group:

  * Aged 18 to 70 years, male or female.
  * Meets the diagnostic criteria for moderate to severe mixed dry eye according to the Expert Consensus on Dry Eye (2020), including:
  * At least one subjective symptom (e.g., dryness, foreign body sensation, burning, fatigue, discomfort, redness, or vision fluctuation).
  * Fluorescein tear film break-up time (FBUT) ≤ 5 seconds.
  * Willing and able to actively cooperate with the prescribed course of standard dry eye medications and ocular surface microbiota transplantation therapy for the study duration.
  * Voluntarily agrees to participate and signs the informed consent form.
* Healthy Donor Group:

  * A family member of a participating subject.
  * Aged 18 to 50 years.
  * Normal ocular surface structure and function, with no ocular diseases or related symptoms, and good visual function.

Exclusion Criteria:

* Dry Eye Patient Group:

  * History of systemic chronic diseases (e.g., uncontrolled diabetes, autoimmune disorders).
  * Current or past history of eyelid abnormalities, conjunctival disease, or lacrimal duct obstruction.
  * History of any ocular surgery or regular wear of corneal contact lenses.
  * Active infection in the eye(s) or any other part of the body.
  * History of multiple episodes of viral keratitis or presence of significant neurotrophic keratitis.
  * Any other condition deemed by the investigator to be unsuitable for participation.
* Healthy Donor Group:

  * Known infectious diseases (e.g., HIV, Hepatitis B).
  * Signs or symptoms suggestive of active ocular surface infection or other viral infections.
  * Current or past history of eyelid, conjunctival, or lacrimal duct diseases.
  * Use of systemic medications (including antibiotics), traditional Chinese herbal medicine, or probiotic supplements within 1 month prior to screening.
  * Pregnancy, lactation, or any other condition that may potentially affect the study outcomes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Score on the Visual Analog Scale (VAS) for Ocular Discomfort | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  The severity of ocular discomfort (e.g., dryness, pain) is assessed using a 100-mm Visual Analog Scale (VAS). Participants mark their level of discomfort on a line from 0 mm ("no discomfort") to 100 mm ("worst imaginable discomfort"). The score is the distance measured in millimeters (mm). A higher score indicates more severe symptoms (worse outcome).

SECONDARY OUTCOMES:
Corneal Fluorescein Staining Score (using the NEI scale) | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  Corneal epithelial damage is assessed by fluorescein staining and graded according to the National Eye Institute (NEI) scale. Each of the five corneal areas is scored from 0 (no staining) to 3 (severe confluent staining). The total score is the sum of all areas, ranging from 0 to 15. A higher score indicates more severe corneal damage (worse outcome).
Change in conjunctival sac microbiota composition assessed by 16S rRNA gene sequencing | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  Microbiota from conjunctival sac swab samples is analyzed using 16S rRNA gene sequencing. Key outcomes include: 1) Alpha diversity change (Shannon Index, unitless), where a higher index indicates greater microbial richness and evenness; 2) Beta diversity change (Weighted UniFrac distance, unitless), measuring compositional shifts between samples; and 3) Change in relative abundance (%) of specific bacterial taxa (e.g., *Corynebacterium*, *Pseudomonas*).
Result of Schirmer I Test (without anesthesia) | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  Tear production is measured by the Schirmer I test (without topical anesthesia). A standardized paper strip is placed in the lateral canthus for 5 minutes. The length of wetting is measured in millimeters (mm). A lower value indicates reduced tear secretion.
Tear Film Break-Up Time (TBUT) | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  Tear film stability is assessed by measuring the tear film break-up time (TBUT). After instillation of fluorescein, the time interval between the last complete blink and the first appearance of a dry spot on the cornea is recorded in seconds (s). A shorter time indicates greater tear film instability.
Score on the Ocular Surface Disease Index (OSDI) Questionnaire | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  Symptoms related to dry eye disease and their impact on vision-related function are assessed using the Ocular Surface Disease Index (OSDI) questionnaire. The total score ranges from 0 to 100, calculated based on responses to 12 items. A higher score indicates more severe disability (worse outcome).
Change in tear fluid inflammatory cytokine levels | At baseline (pre-intervention), and at 1 week, 2 weeks, and 4 weeks post-intervention.
  Levels of inflammatory cytokines in tear fluid samples are measured using a multiplex immunoassay (e.g., Luminex assay or ELISA). The concentration of specific cytokines (e.g., IL-1β, IL-6, IL-8, TNF-α) is reported in picograms per milliliter (pg/mL). An increase in concentration indicates a higher level of inflammation (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Yifeng Yu, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided